CLINICAL TRIAL: NCT07254078
Title: Registry of Patients With Chronic Thromboembolic Pulmonary Hypertension in Russia: Determinants of Long-term Outcomes in Real Clinical Practice
Brief Title: Registry of Patients With chrOnic thromboemboLic Pulmonary hypErTension
Acronym: POLET
Status: Recruiting | Type: Observational
Sponsor: Irina E. Chazova (Other Government)
Responsible Party: Sponsor-Investigator, Irina E. Chazova, D. Sci. (Med.), Acad. RAS, Prof., Deputy Director General for Scientific and Expert Work, FSBI NATIONAL MEDICAL RESEARCH CENTRE OF CARDIOLOGY NAMED AFTER ACADEMICIAN E.I.CHAZOV of the Ministry of Health of the Russian Federation, National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Organization: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Other Study IDs: 313
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: CTEPH; registry; PEA; BPA; PAH-specific therapy; survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Pulmonary endarterectomy — A surgical procedure to remove chronic blood clots from the pulmonary arteries
  Other Names: PEA; PTE; Pulmonary thromboendarterectomy
Procedure: Balloon pulmonary angioplasty — A minimally invasive procedure used to treat chronic thromboembolic pulmonary hypertension by dilatating narrowed pulmonary arteries and improving blood flow to the lungs
  Other Names: BPA
Drug: Pulmonary hypertension-specific therapy — Medical treatment with any PH-specific drugs
  Other Names: PH-specific therapy; PH-Targeted Medical Therapy

SUMMARY:
The goal of this observational study is to gather information on background, medical history, symptoms and physical condition, treatment options of people with chronic thromboembolic pulmonary hypertension in real clinical practice in Russia.

The main question it aims to answer is:

Which factors most influence the prognosis of participants?

DETAILED DESCRIPTION:
Data from international CTEPH registries indicate variable utilization rates of available treatment options. Considering the presence of national specificities in the management of CTEPH patients, coupled with the relatively low prevalence of the disease, which poses challenges for data accumulation and research, new registry POLET (Registry of Patients with chrOnic thombomboLic pumonary hypErTension) is established to investigate CTEPH patients in real-world clinical practice.

Registry Aim:

To investigate the prognosis of patients with chronic thromboembolic pulmonary hypertension based on demographic, anamnestic, clinical characteristics, and treatment regimens.

Registry Objectives:

To describe the key demographic, anamnestic, and clinical characteristics of CTEPH patients in Russia.

To identify factors influencing the frequency of hospitalizations due to clinical deterioration in CTEPH patients.

To determine the impact of anamnestic data and treatment regimens on patient prognosis (time to clinical deterioration/death).

To determine the impact of demographic and clinical characteristics on patient survival and prognosis (time to clinical deterioration/death).

Currently, preliminary retrospective data have been collected on 300 CTEPH patients, each with 1 to 15 hospitalizations at the National Medical Research Center of Cardiology named after Academician E.I. Chazov of the Ministry of Health of Russia from 2012-2024, and who are eligible for inclusion in the registry. 200 patients will be enrolled prospectively.

The following data to be extracted from electronic medical records:

Medical History Data; Clinical Characteristics and Results of Investigations and Treatments During Each Patient Hospitalization; Operability Assessment Results; PAH-Specific Therapy, Anticoagulant Therapy, Supportive Therapy: Therapy Adjustment, Doses, Presence of Side Effects; Details of Pulmonary endarterectomy; Details of BPA performed; Patient outcomes including survival. Statistical data processing will be performed using RStudio and the R programming language. Missing data will be handled with imputation approach.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a confirmed diagnosis of CTEPH

Exclusion Criteria:

* Presence of pulmonary hypertension of a different etiology than CTEPH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: operable CTEPH, non-operable CTEPH
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2035-05-01 (Estimated); Study Completion 2035-05-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Up to 5 years

SECONDARY OUTCOMES:
All-cause mortality | Up to 10 years
Change in distance in 6-minute walk test | 1 year
Change in mPAP | 1 year
  mPAP assesed during right heart catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center of Cardiology after academician E.I. Chazov, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No